CLINICAL TRIAL: NCT04705506
Title: Effect of Gemigliptin on Biomarkers of Kidney Injury and Vascular Calcification in Diabetic Nephropathy: A Randomized Controlled Trial
Brief Title: Gemigliptin and Biomarkers of Kidney Injury and Vascular Calcification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 186/60
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Nephropathies
Keywords: Gemigliptin; Diabetic Nephropathy; Acute Kidney Injury; Vascular Calcification
MeSH Terms: conditions — Diabetic Nephropathies; Acute Kidney Injury; Vascular Calcification | interventions — LC15-0444

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, randomized, placebo-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemigliptin group (Experimental): The participants will receive gemigliptin 50 mg daily
  Interventions: Drug: Gemigliptin
- Control (Placebo Comparator): The control received standard care of diabetes
  Interventions: Drug: Gemigliptin

INTERVENTIONS:
Drug: Gemigliptin — We collected baseline data from all participants for demographic characteristics,comorbid conditions and biochemistry indexes.The biomarkers for vascular calcification and renal injury were collected.Baseline CAC score and CAVI were done.The patients then were randomized into 2 groups: Group 1 received gemigliptin 50 mg /day for 6 months in addition to standard treatment ,Group 2 will have standard treatment for diabetes mellitus (DM) and chronic kidney disease (CKD).The patients will be followed up every eight weeks.Fasting plasma glucose ,BUN creatinine and 24 hour urine protein were measured at each study visit.Patients were scheduled for follow-up visits at months 2,4,and 6.After 6 months ,all the blood tests,CAC score and CAVI will be done again.
  Other Names: Treatment group

SUMMARY:
Dipeptidyl peptidase-4 (DPP-4) inhibitors improve glycemic control and contain pleiotropic actions on kidney injury, albuminuria and vascular inflammation especially in animal models. We plan to evaluate the efficacy of potent DPP4-inhibitors (gemigliptin) in response to these aspects in diabetic nephropathy patients.

DETAILED DESCRIPTION:
This is a multi-center, prospective, randomized, placebo-controlled trial. A total of 201 participants were enrolled and randomly assigned to gemigliptin 50 mg daily and standard care of diabetes mellitus for 6 months. The changes of coronary calcium score (CAC score), cardio-ankle vascular index (CAVI), estimated glomerular filtration rate (GFR), markers of vascular calcification and markers of tubular renal injury were evaluated at baseline and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD stage 1-3 (eGFR 15-60 ml/min/1.73mL)
* Non-insulin dependent diabetes mellitus , blood glucose level 30-250 mg/dL
* Had clinical features compatible with diabetic nephropathy (urine micro albuminuria > 30 g/g creatinine or has evidence of diabetic retinopathy

Exclusion Criteria:

* History of allergy to DPP4-inhibitor
* Concurrent infectious disease
* Inflammatory diseases
* Post kidney transplantation
* Receiving cinacalcet, bisphosphonate ,previously treated with DPP4-Inhibitors and sodium-glucose cotransporter-2 inhibitor (SGLT2-i).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Markers of renal injury | 6 months
  urine NGAL/Cr,urine Kim-1/Cr,urine LFABP/Cr (pg/mL)
Markers of vascular calcification | 6 months
  serum bone alkaline phosphatase(pg/mL),osteopontin (pg/mL)
Markers of renal injury | 6 months
  Protienuria (mg/day)
Markers of renal injury | 6 months
  eGFR (mL/min/1.73m2)
Markers of vascular calcification | 6 months
  Reactive oxygen species (ng/mL)
Markers of vascular calcification | 6 months
  CAVI,CAC score(unit) ,CAVI normal less than8 ,CAC score normal less than 100

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvanich, M.D., Principal Investigator — Navamindradhiraj University
Locations (3):
- Thailand (3):
  - Faculty of Medicine ,Vajira Hospital, Bangkok
  - 2 Division of Nephrology,Department of Medicine Pramongkutklao Hospital and College of Medicine,Thailand, Bangkok
  - Department of Medicine,Police General Hospital,Thailand, Bangkok

REFERENCES:
- [Derived] Trakarnvanich T, Satirapoj B, Suraamornkul S, Chirananthavat T, Sanpatchayapong A, Claimon T. Effect of Dipeptidyl Peptidase-4 (DPP-4) Inhibition on Biomarkers of Kidney Injury and Vascular Calcification in Diabetic Kidney Disease: A Randomized Controlled Trial. J Diabetes Res. 2021 Oct 16;2021:7382620. doi: 10.1155/2021/7382620. eCollection 2021. PMID 34697593